CLINICAL TRIAL: NCT01504113
Title: The Impact of Targeted Therapy on Microorganism in Patients With Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201106079RC
Record Dates: First submitted 2011-08-03; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-07

CONDITIONS: Psoriasis
Keywords: Target therapy; Biologics; Psoriasis; Latent virus; Human papillomaviruses; Cytomegalovirus; Epstein-Barr virus; Tumor necrosis factor
MeSH Terms: conditions — Psoriasis; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and skin scales

GROUPS / COHORTS (3):
- Study 1 goup: Patients who are planned to receive targeted agents
- Study 2 case group: Patients who have received targeted therapy
- study 2 control group: Psoriasis patients without target therapy

SUMMARY:
Background:

Psoriasis is a chronic, immunologically-mediated, inflammatory skin disease and targeted therapies e.g. tumor necrosis factor (TNF)-α and TH-17 antagonists have become increasing important agents in the management of psoriasis. TNF, interleukin-17 (IL-17) and TH-17 play major roles in defense against infection. Large-scaled clinical trials and post-marking surveillance had shown these agents may increase susceptibility to infections. Most studies evaluate the reactivation of tuberculosis but the influence of targeted therapies on the viral infection has not been extensively investigated.

TNF-α has been shown to contribute to the killing of cytomegalovirus (CMV)- and human papillomaviruses (HPV)-infected cells. Additionally, recent studies have shown a high prevalence of HPV DNA in psoriatic skin and increased HPV5 antibodies in patients with psoriasis. The prevalence of HPV in the skin was also affected by therapeutic modalities, such as psoralen-ultraviolet A (PUVA). Several case reports in which CMV, Epstein-Barr virus (EBV) and HPV infection complicated therapy with TNF-α antagonists have been reported. However, the study investigated the effect of TNF-α antagonists and other biologics on reactivation of latent viruses is limited. Only two studies investigated the short-term effect of infliximab on reaction of herpesviruses in patients of rheumatoid arthritis and Crohn's disease. The high prevalence of combination use of immunosuppressants, such as methotrexate alongside with TNF-α antagonists in these patients is different from patients with psoriasis. Additionally, various bacterium and fungi, such as Staphylococcus aureus, Malassezia are associated with provocation and/or exacerbation of psoriasis and recent studies had shown IL-17 is essential for the immune response to common fungus Candida albicans.

Aim:

The aim of this study is to prospectively investigate the effect of target therapies (TNF-α, TH-17 antagonist, IL-17 antagonists, tofacitinib and apremilast) on the activation of viruses, including CMV, EBV and HPV and the impact of biologics on the prevalence of surface colonization of microorganism, including HPV, bacteria and fungi, in patients with psoriasis.

Methods and procedures:

Our project consists of two related study. The first (Study 1), a prospective observational study, included patients with psoriasis who are going to undergo biologics therapy, the viral loads of CMV and EBV, HPV DNA detection in eyebrow hairs and skin scales, and bacterial, fungal cultures from skin scales were performed before the initiation, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. This part of our project is to investigate the dynamic effect of biologics on the microorganisms in patients with psoriasis. The second part (Study 2), a case control study, recruits psoriasis patients who have started target therapies, they receive the sampling of blood, eyebrow hairs and skin scales for CMV, EBV and HPV investigations when they are enrolled. Control group compromised of age-and disease severity-matched psoriasis patients who are not treating with target therapies or other systemic antipsoriatic agents. Comparison of the prevalence of latent virus, virus reactivation, bacteria and fungi skin colonization between psoriasis patients who are treating with and without target therapies is performed. The aim of study 2 was to assess any difference of the status of latent virus or microorganism colonization in skins between psoriasis patients treated with and without target therapies.

DETAILED DESCRIPTION:
Introduction As numerous studies have identified TNF-α, TH-17 and IL-17 as particularly major roles governing the inflammatory cascade in psoriasis, target therapies, including TNF-α and TH-17 antagonists, have represented major breakthrough in the treatment of psoriasis. It is well known that TNF-α plays an important role in the immune response to viral infections, which is attributed to direct inhibition of viral replication, killing of virally infected cells, induction of FasL-dependent CD8+ T-lymphocyte effector pathways through TNF/TNF receptor 2 interaction and promote inflammatory response indirectly.Additionally, it has been shown that treatment with TNF-α antagonists is associated increased viral replication in virus-inoculated rats, progressive loss of CD4+ and CD8+ T cells and decreased level of TNF-α and interferon. A transient decreased T cell responsiveness was also observed in some patients treated with TNF-α antagonists.10 TNF-α can inhibit CMV production in certain cell types and the CMV major immediate early promoter is inhibited by TNF-α. Increased TNF production has been reported during CMV infection, which also displays anti-CMV activity in vitro.

TNF-α is also involved in direct control of HPV infection by induction of apoptosis of HPV-infected cells, arresting growth of HPV-infected keratinocytes and down-regulation of HPV-gene transcription, stimulation of inflammatory response and up-regulation of HLA class I components in antigen-presenting cells. E6 protein of HPV-16 is known to directly bind to TNF receptor 1 and abrogate TNF-induced apoptosis of the host cells. Recent studies have shown a high prevalence of HPV DNA in psoriatic skin and increased HPV5 antibodies in patients with psoriasis. It seems that psoriatic skin may be specifically permissive for HPV. Increased pap smear abnormalities has been observed in patients with inflammatory bowel diseases receiving TNF-α antagonists. However, the specific effects of anti-TNF therapy on HPV carriage and HPV-associated disease remain unknown.

Epstein-Barr virus (EBV) is associated with several B-cell and epithelial-cell malignancies, especially in patients under the immunosuppressive treatment. Increased risk of lymphoproliferative disorders in patients treated with TNF-α antagonists has been addressed. Case reports of EBV-associated lymphoproliferative diseases that regressed after withdrawal of anti-TNF-α drugs had been also described. Thus, the concern of the increased risk at least in part caused by immunosuppression of anti-TNF therapy, which may cause a consecutive EBV reactivation, emerged but was not proven yet.

Anti-TNF-α drugs, including monoclonal antibody against TNF-α (infliximab and adalimumab) and soluble TNF receptor (etanercept), are recognized as a risk factor for opportunistic infections. A recent study demonstrated a higher risk of opportunistic infections for patients receiving adalimumab than etanercept, with a 10- to 17-fold differences in risk. However, most knowledge of latent viral reactivation during anti-TNF treatment has come from studies of patients with inflammatory bowel disease and rheumatoid arthritis. Moreover, these studies mainly focus on herpesviruses and viral hepatitis. Several case reports in which EBV, CMV,and HPV infection complicated therapy with TNF-α antagonists in patients with psoriasis have also been reported.

IL-17 is a proinflammatory cytokine that is produced by a variety of cells, including a newly identified subset of activated CD4+ T cells (Th17 cells), γδT cells, CD8+ cells and NKT cells. There is evidence to support a protective role for IL-17 in the host defense against extracellular bacterial infections, including Klebsiella pneumonia,38 Bacteroides fragilis and Escherichia coli. A recent study also showed IL-17 is essential for human immunity against common fungus Candida albicans.

Various bacteria and fungi are reported to be associated with provocation and/or exacerbation of psoriasis. The strongest evidence exists for the induction of guttate psoriasis by a preceding tonsilar Streptococcus pyogenes infection. Balci et al also found significant higher rates of Staphylococcus aureus colonization in lesional skin and nares of the patients with psoriasis than healthy controls. They also suggested a significant relationship between PASI scores and both S. aureus cultivation and toxin production in lesional skin of the patients with psoriasis.

However, the studies investigating the impact of TNF-α, TH-17, IL-17 antagonists and other targeted agents in patients with psoriasis are limited.

Aim： In Taiwan, the seropositive rate of CMV is approximately 50% for school age children and more than 90% for adults. EBV causes a persistent infection of B lymphocytes in more than 90% of the adult population worldwide.46 Thus, the importance of investigating the influence of target therapies on the latent viruses and other microorganisms can't be overemphasized. The aim of this study is to prospectively investigate the effect of TNF-α, TH-17 and IL-17 antagonists administration on the activation of viruses, including CMV, EBV and HPV and the impact of biologics on the prevalence of surface colonization of microorganism, including HPV, bacteria and fungi, in patients with psoriasis. The microbial effect of novel targeted agents, like tofacitinib, secukinumab and apremilast, will also be studied.

Methods Patients Characteristics and Study Schedule We include patients with psoriasis who will receive and who are currently on TNF-α (etanercept and adalimumab) for psoriasis, in a tertiary referral centre in northern Taiwan (National Taiwan University Hospital (NTUH)) between 2011 and 2015. We also include patients who have signed informed consent to use or participate in the clinical trials and are currently using the target therapies of ustekinumab, secukinumab, tofacitinib (CP690,550), and apremilast. These clinical trials are approved by the Research Ethics Committee of the NTUH (NTUH-REC: ustekinumab, 200806022M; secukinumab, 201104022MA; tofacitinib, 201012013MA; apremilast, 201010022M). Patients themselves or their guardians have signed informed consent for the study protocols of these new drugs before entrance to this study. All the participants of our study or their guardians also need to sign another informed consent of this study, which is approved by the Research Ethics Committee of the NTUH (NTUH-REC No: 201106079RC).

This project consists of two related studies:

Study 1

1. Patients who are planned to receive targeted agents:

   This prospective, observational study includes psoriasis patients who are going to receive targeted agents. After enrollment, CMV and EBV IgG are checked. Patients undergo the sampling of blood, eyebrow hairs and skin scales before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. Blood samples are sent to check viral load, and CMV and EBV viral load are determined by real-time PCR. Bacterial, fungal cultures and HPV DNA detection of skin scales are also performed. HPV typing is determined by genechip and semi-quantitative measurement of HPV viral load is done. Demographic data and the activity parameters of the psoriasis, such as psoriasis area and severity index (PASI), are collected at baseline and each study visit. The aim of this study is to investigate the dynamic effect of target therapies administration on the microorganisms, including CMV, EBV, HPV, bacteria and fungi in patients with psoriasis.

   Study 2
2. Patients who have received targeted therapy The second part of our project, a case-control study, includes psoriasis patients who have received targeted agents for more than 3 months. We also recruit age-and disease severity-matched psoriasis patients who are not treating with targeted agents or other systemic antipsoriatic agents as a control group. Likewise, after enrollment, CMV and EBV IgG are checked. HPV detection, bacterial, fungal cultures of the skin scales were done. Comparison of the prevalence of latent virus, virus reactivation, bacteria and fungi skin colonization between psoriasis patients who are treating with and without target therapies is performed.

Additionally, the microorganism examinations are repeated again 12 weeks after the discontinuation of target therapies. The dynamic changes of viral serology, bacterial and fungal cultivation data after stopping target therapies are analyzed.

The aim of this part of our study was to assess any difference of the status of latent virus or microorganism colonization in skins between psoriasis patients treated with and without target therapies.

Scale sampling on the nonlesional skins for HPV The sampling areas will be first cleaned with Hibitane and gentlely taped with adhesive tapes to remove surface contamination. Then a superficial skin scraping is taken from the head and neck areas, as far as possible from any psoriatic plaques, using a fine sandpaper to abrade the stratum corneum and collecting the debris for HPV detection.

Cultivation of bacteria and fungi on the skin folds After clearing sampling areas with Hibitane, skin swab samples are taken from skin folds, including retroauricular areas, inguinal or axillary areas, by using a sterile cotton swab dipped in double-distilled water and then a gentle swabbing of the skin.

Hair sampling for HPV Eyebrows are plucked with new tweezers used for each subject. Only hairs containing intact hair follicles are collected for HPV studies.

Determination of viral loads

Quantitative PCR for CMV and EBV viral load Whole blood specimens were stored at - 80 ◦C before testing. DNA was extracted from 400μL of sample with the MagNA Pure Compact Nucleic Acid Isolation kit I using the MagNA Pure Compact Instrument (Roche Diagnostics). The volume of solution was 100μL. Viral DNAs were then amplified using the "in-house" real-time PCR assays implemented in the laboratory for virological diagnosis. For CMV, real-time PCR assays based on hydrolysis probe technology were used, as described previously.48 For EBV, the "in-house"real-time PCR assay using hybridization probes was carried out, as reported previously.49 CMV amplification was performed on the ABI PRISM® 7500 (Applied Biosystems, Courtaboeuf, France) using the following cycle parameters: 2 min at 50 ◦C and 10 min at 95 ◦C, followed by 45 cycles each consisting of 15 s at 95 ◦C and 1 min at 60 ◦C (ramprates of 0.8 ◦C/s up and 1.6 ◦C/s down; 9600 emulation mode). EBV assay was carried out on the LightCycler® 1.5 (LC1.5; Roche Diagnostics). EBV assay was performed with the following cycle parameters: 1 min at 50 ◦C and 8 min at 95 ◦C, followed by 45 cycles each consisting of 10 s at 95 ◦C, 15 s at 58 ◦C and 15 s at 72 ◦C, and a cooling step of 1 min at 40 ◦C (ramp rate of 20 ◦C/s). Real-time PCR assays were performed in parallel on the LC480, after slight adaptations from the initial protocols. Ten microliters of extracted DNA were amplified in 25μL of mixture containing 1 × LightCycler® 480 Probes Master, 200 nM forward primer, 200 nM reverse primer, 100 nM hydrolysis probe, 0.38 units uracil-N-glycosylase (Invitrogen, Cergy-Pontoise, France). For EBV, the hybridization probe labeled with LC-Red 640 was used as a FAM-labeled hydrolysis probe.49 The sequences of all primers and probes used in LC480 protocols are indicated in Table 1. Cycling conditions on LC480 were as follows: 2 min at 50 ◦C and 10 min at 95 ◦C, followed by 45 cycles each consisting of 15 s at 95 ◦C and 40 s at 60 ◦C, and a cooling step of 30 s at 40 ◦C (ramp rate of 4.4 ◦C/s). For CMV and EBV assays, quantitation was achieved with a standard curve generated from 10-fold serial dilutions of viral DNA extracted from infected cell cultures and quantified using a plasmid. In order to detect potential PCR inhibitors, all DNA extracts were tested undiluted and at a dilution of 1:10. Results were expressed logarithmically (viral copy number/mL). Given the extraction dilution, the sensitivity threshold was 1.4 logs for all assays.

HPV genotyping and semiquantitative HPV viral load The HPV genechip (Easychip HPV Genotyping Array, King Car, Taipei, Taiwan) will offer an revert-blot hybridization to detect 39 subtypes of HPV DNA (6, 11, 16, 18, 26, 31, 32, 33, 35, 37, 39, 42, 43, 44, 45, 51, 52, 53, 54, 55, 56, 58, 59, 61, 62, 66, 67, 68, 69, 70, 72, 74, 82, CP8061, CP8304, L1AE5, MM4, MM7, and MM8) in a single reaction, as reported by Huang et al. The nested multiplex PCR products of L1 region of HPV of each specimen will be hybridized with a genechip. The other set of nested PCR will be also performed for skin typed HPV which consisted of FAP59/64 and Fap6319R/6085F and DNA sequencing analysis.will be performed for the product to rule out the presence of coinfection. The genechip is able to detect multiple infection and the skin-directed PCR sequencing can only detect one serotype of HPV at one time. Internal Control for extracting of human-genomic DNA

1. . GAPDH, gap-1/gap-2 (ca. ~341 bp)
2. . Beta-globin, KW42/KW29 (ca. ~510 bp)
3. . Beta-globin, KC03/KC04 (ca. ~110 bp)
4. . Beta-globin, KC03/KC05 (ca. ~150 bp)

Strategy of mucosal HPV detection:

Primers mDeAV1 5'-CGTCCM*ARRGGAWACTGATC-3' mDeAV2 5'-GCMCAGGGWCATAAYAATGG-3'-Biotin GAP1: 5'-CCAACTTTCCCGCCTCTCAGC-3' GAP2: 5'-AAAACCGCTAGTAGCCGGGCC-3' KW29: 5'-GGTTGGCCAATCTACTCCCAGG-3' KW42: 5'-GCTCACTCAGTGTGGCAAAG-3'

For the detection of skin typed HPV, the other sets of nested PCR primer will be used as:

FAP59：5'-TAACWGTIGGICAYCCWTATT-3') FAP64：5'-CCWATATCWVHCATITCICCATC-3') FAP6085F：CCWGATCCHAATMRRTTGC FAP6319R：ACATTTGGGGGAAAAATTGTTTDGGRTCAA The amount of HPV DNA in the specimen was determined by semiquantitative method. Luminescence signal strengths in relative light units (RLU) of the specimen were compared with standard positive controls (RLU/PC).

ELIGIBILITY:
Study 1

Inclusion Criteria:

* Clinical diagnosis of psoriasis/psoriatic arthritis and are going o receive target therapies in the near future
* Age more than 20 years old
* Will receive target therapies for psoriasis/psoriatic arthritis
* Willing to receive blood, hair and skin scale sampling

Exclusion Criteria:

* Pregnancy
* Not candidates for topical therapies, such as :

Active tuberculosis or HIV, human papillomaviruses, cytomegalovirus infection, Epstein-Barr virus infection Evidence of latent tuberculosis but refuse to receive isoniazid prophylaxis Have malignancy required for chemotherapy or radiotherapy Active uncontrolled hepatitis -Have received phototherapy, systemic immunosuppressants or target therapies within 14, 30, 84 days prior to enrollment, respectively Study 2 (case group)

Inclusion Criteria:

* Clinical diagnosis of psoriasis/psoriatic arthritis
* Age more than years old
* Have received target therapies for more than 3 months
* willing to receive blood, hair and skin scale sampling

Exclusion Criteria:

* Pregnancy
* Not candidates for topical therapies, such as :

Active tuberculosis or HIV, human papillomaviruses, cytomegalovirus infection, Epstein-Barr virus infection Evidence of latent tuberculosis but refuse to receive isoniazid prophylaxis Have malignancy required for chemotherapy or radiotherapy Active uncontrolled hepatitis

-Have received phototherapy, or systemic immunosuppressants within 14 and 30 days prior to enrollment,respectively Study 2 (control group)

Inclusion Criteria:

* Clinical diagnosis of psoriasis/psoriatic arthritis and are going o receive target therapies in the near future
* Age more than 20 years old
* Willing to receive blood, hair and skin scale sampling
* Without phototherapy, systemic immunosuppressants or target therapies within 84 days prior to enrollment, respectively

Exclusion Criteria:

* Pregnancy
* Have received phototherapy within 30 days prior to enrollment

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include patients with psoriasis who will receive and who are currently on target therapies,such as TNF-α, TH17,and IL-17 antagonists for psoriasis, in a tertiary referral centre in northern Taiwan (National Taiwan University Hospital (NTUH)) between 2011 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in viral loads of human papillomaviruses virus during and after target therapy | before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies
  Study 1:The sampling of eyebrow hairs and skin scales before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. Study 2: The same above mentioned microorganisms exams were done at enrollment and repeated again 12 weeks after the discontinuation of therapies. Comparison of the prevalence of latent virus and changes from baseline in viral load of human papillomaviruses virus between psoriasis patients who are treating with and without target therapies is performed.
Changes from baseline in viral loads of cytomegalovirus during and after target therapy | before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies
  Study 1:The sampling of blood before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. Study 2: The same above mentioned microorganisms exams were done at enrollment and repeated again 12 weeks after the discontinuation of therapies. Comparison of the prevalence of latent virus, and changes from baseline in viral load of cytomegalovirus between psoriasis patients who are treating with and without target therapies is performed.
Changes from baseline in viral loads of Epstein-Barr virus during and after target therapy | before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies
  Study 1:The sampling of blood before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. Study 2: The same above mentioned microorganisms exams were done at enrollment and repeated again 12 weeks after the discontinuation of therapies. Comparison of the prevalence of latent virus, and changes from baseline in viral load of Epstein-Barr virus between psoriasis patients who are treating with and without target therapies is performed.

SECONDARY OUTCOMES:
Changes from baseline in the prevalence of bacterial and fungal skin colonization during and after target therapy | before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies.
  Study 1:The sampling of skin scales before the initiation of biologics therapy, 12 and 24 weeks after initiation of the target therapies, 12 weeks after discontinuation of target therapies. Study 2: The same above mentioned microorganisms exams were done at enrollment and repeated again 12 weeks after the discontinuation of therapies. Comparison of the prevalence of bacteria and fungi skin colonization between psoriasis patients who are treating with and without target therapies is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Tsen-Fang Tsai, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Dermatology department, Taipei, Taiwan